CLINICAL TRIAL: NCT01792622
Title: Patient Reported Outcomes in Pulmonary Arterial Hypertension
Acronym: PROPAH
Status: Withdrawn | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: University of Chicago (Other); Mayo Clinic (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481296
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Instrument Development; Patient Reported Outcomes; Pulmonary Arterial Hypertension.
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase I Patient Interviews: Indepth interviews will be completed with approximately 15 patients.
  Interventions: Other: Interview
- Phase II Patient Questionnaire: Patients will be asked to provide subjective ratings of their experience on a questionnaire developed from the responses from Phase I
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Interview — Patients will be interviewed to provide descriptive information about their experience as a treated patient with pulmonary arterial hypertension. The interviews will be given one time for approximately 1 hour.
  Groups: Phase I Patient Interviews
Other: Questionnaire — Patients will be asked to provide subjective ratings of their experience on a questionnaire developed from the responses from Phase I. The questionnaire will be given one time for approximately 1 hour.
  Groups: Phase II Patient Questionnaire

SUMMARY:
Develop a brief, new, patient reported outcome instrument that is valid for use in clinical practice and clinical trials.

DETAILED DESCRIPTION:
This study will use the Clinical Impact Method to develop a patient reported outcome for use in patients with pulmonary arterial hypertension Clinical personnel at the study sites will approach and discuss possible participation in Phase I and II of the study with subjects from the existing pool of patients currently receiving usual and customary care at the site.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent
* Subjects aged >=18 who have documented PAH
* Speak English
* Subjects who provide written informed consent to participate in the study before being screened for the study.

Exclusion Criteria:

* Patients with non-PAH Pulmonary Hypertension
* Physical inability to complete the interview process
* Subjects who are currently enrolled in an experimental drug study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for the study will be a composite symptom score derived from items in the instrument. | Patients in Phase 1 and 2 shall be engaged in the study for approximately one hour's time; Phase 1 will take 3 to 6 weeks, and Phase 2 will proceed until sufficient sample size is obtained (saturation); we anticipate completion by September 2013.
  Composite symptom score shall be derived from the actual items selected as a result of Phase 2.
  The final scoring logarithm shall provide a score for each dimension, as well as an anxiety/concern scale derived from single items from each of the dimensions, and a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481296&StudyName=Patient%20Reported%20Outcomes%20in%20Pulmonary%20Arterial%20Hypertension